CLINICAL TRIAL: NCT03086824
Title: A Safety Evaluation of MR-guided Focused Ultrasound Treatment for Palliative Pain Control of Bone Metastases
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Jo-Ting Tsai, Doctor of Philosophy(Ph.D.)/Director, Department of Radiation Oncology, Taipei Medical University - Shuang Ho Hospital, New Taipei, Taiwan, Taipei Medical University Shuang Ho Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMU-SHH-2014-001
Record Dates: First submitted 2016-12-07; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Magnetic Resonance Guided Interventional Procedures
Keywords: Bone Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRgFUS (Experimental): Patients with painful bone metastases receiving magnetic resonance-guided focused ultrasound treatment.
  Interventions: Device: magnetic resonance-guided focused ultrasound

INTERVENTIONS:
Device: magnetic resonance-guided focused ultrasound

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of subjects receiving MR-guided Focused Ultrasound (MRgFUS) treatment for painful bone metastases. This study will evaluate treatment response and clinically significant adverse events. Other relevant data may be documented as well.

DETAILED DESCRIPTION:
This proposed study will be performed in full compliance with all applicable privacy rules and regulations, and their implementations at participating site(s). All subjects planned to undergo the MRgFUS procedure at Taipei Medical University Hospital will be offered informed consent so they can be included in this Study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 20 and older.
2. Patients who are able and willing to give consent and able to attend all study visits.
3. Patients who are suffering from symptoms of bone metastases: Patients who have received radiation without adequate relief from metastatic bone pain as determined by the patient and treating physician, those for whom their treating physician would not prescribe radiation or additional radiation treatments, and those patients who refuse additional radiation therapy.
4. Patient with NRS (0-10 scale) pain score ≥ 4 irrespective of medication.
5. Targeted bone/tumor interface are ExAblate device accessible and are located in ribs, extremities (excluding joints), pelvis, shoulders and in the posterior aspects of the following spinal vertebra: Lumbar vertebra (L3-L5), Sacral vertebra (S1-S5).
6. Patient whose targeted lesion is on bone and the interface between the bone and lesion is deeper than 10-mm from the skin.
7. Targeted (treated) tumor clearly visible by non-contrast MRI, and ExAblate MRgFUS device accessible.
8. Patients on ongoing chemotherapy regimen at the time of eligibility: 1) with same chemotherapy regimen (as documented from patient medical dossier, 2) worst pain NRS still ≥ 4, and 3) do NOT plan to initiate a new chemotherapy for pain palliation should be eligible for the study. Note: Planned multiple courses of chemotherapy are not considered New Chemotherapy.
9. No radiation therapy to targeted (most painful) lesion in the past two weeks.
10. Bisphosphonate intake should remain stable throughout the study duration. -

Exclusion Criteria:

1. Patients who either Need surgical stabilization of the affected bony structure or Targeted tumor is at an impending fracture site or Surgical stabilization of tumor site with metallic hardware.
2. KPS (Karnofsky performance scale) Score < 60.
3. Unable to communicate sensations during the ExAblate treatment.
4. Target (treated) tumor is less then 10-mm from nerve bundles, bowels or bladder.
5. Patients with acute medical condition (e.g., pneumonia, sepsis) that is expected to hinder them from completing this study.
6. Severe cerebrovascular disease (multiple CVA or CVA within 6 months).
7. Patients with unstable cardiac status (e.g. unstable angina pectoris, myocardial infarction within 6 months, congestive heart failure NYHA Class IV, on arrhythmic drugs).
8. Severe hypertension (diastolic BP > 100 mmHg on medication).
9. Patients on dialysis.
10. Patients with standard contraindications for MRI or MRI contrast agents. -

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-12-12 (Actual); Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Treated-related Adverse Events | 12-months

SECONDARY OUTCOMES:
Change from baseline Quality of Life Questionnaire | 1day, 3days, 1-week, 2-weeks, 1-month, 2-months, 3-months, 6-months, 9-months, 12-months
Change from baseline Pain Score | 1day, 3days, 1-week, 2-weeks, 1-month, 2-months, 3-months, 6-months, 9-months, 12-months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Taipei Medical University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes